CLINICAL TRIAL: NCT07061457
Title: Brachial-radial Pressure Gradient Phenomenon in Critically Ill Patients Treated With Vasoactive Agents: an Observational Study
Brief Title: Brachial-radial Pressure Gradient Phenomenon in Critically Ill Patients Treated With Vasoactive Agents
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Wojciech Szczeklik, Professor, Jagiellonian University
Other Study IDs: 118.0043.1.305.2024
Record Dates: First submitted 2025-06-18; First posted 2025-07-11 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-07

CONDITIONS: Circulatory Failure; Shock; Vasopressor Agents; Blood Pressure
Keywords: brachial-to-radial gradient; vasoactive agents; vasopressor; critically ill
MeSH Terms: conditions — Shock; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult critically-ill patients receiving vasoactive agents: Adult critically-ill patients receiving vasoactive agents and undergoing invasive blood pressure monitoring in the radial artery

SUMMARY:
The goal of this observational study is to observe brachial-to-radial pressure gradient in critically-ill patients receiving vasoactive agents. The main questions it aims to answer are:

1. What is the frequency of brachial-to-radial gradient in critically-ill patients receiving vasoactive agents?
2. Is brachial-to-radial gradient greater in patients receiving high doses of vasoactive agents?
3. Is brachial-to-radial gradient associated with worse peripheral perfusion?

DETAILED DESCRIPTION:
Pathological conditions, such as arterial stenosis, use of vasoconstrictive drugs, or massive vasodilatation, can cause significant differences in mean arterial pressure (MAP) in different parts of the arterial system. For example, in the case of stenosis between the brachial and radial arteries, the pressure behind the stenosis is lower than in front of it, which can lead to erroneous conclusions about the actual arterial pressure. The use of vasoconstrictive drugs in patients with circulatory insufficiency can result in reduced peripheral arterial pressure transmission, as evidenced by studies showing lower pressures in the radial artery compared to the femoral artery. Inadequate MAP assessments can lead to excessive use of vasoactive drugs and fluids, increasing the risk of complications such as cardiac ischemia, atrial fibrillation, and renal failure. One method to detect a significant gradient between central MAP (e.g., aorta or femoral artery) and peripheral MAP is non-invasive, oscillometric measurement of MAP on the brachial artery and comparing it to MAP obtained from invasive radial access (known as NIBR-APG). The brachial-radial MAP gradient is highly correlated with the femoral-radial gradient and may be indicative of significantly higher central pressure. The aim of this project is to evaluate the frequency of the brachial-radial gradient phenomenon in patients undergoing vasoconstrictive treatment in intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* adult (>18 years) patients admitted to the ICU
* must be after initial resuscitation
* invasive blood pressure monitoring in the radial artery
* need for vasoactive drug therapy

Exclusion Criteria:

* pregnancy
* pressure transduction across invasive blood pressure circuit deemed to be inadequate
* mechanical circulatory support
* inability to match non-invasive cuff size to the patient's arm
* need for any hemodynamic intervention during performing study's measurements
* patient's decline to have the measurements done

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the intensive care unit, requiring invasive blood pressure monitoring, and undergoing vasoactive therapy.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2025-04-14 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Frequency of significant brachial-to-radial gradient | At baseline (after initial resuscitation). The gradient will be assessed only once, in a cross-sectional manner.
  Frequency of significant brachial-to-radial gradient > 11 mmHg MAP

SECONDARY OUTCOMES:
Determinants of the brachial-to-radial gradient | At baseline (after initial resuscitation). The variables will be collected only once in a cross-sectional manner.
  Odds ratio (OR) of norepinephrine equivalent dose and OR of other potential risk factors (diabetes, age and body surface area) for significant brachial-radial gradient (>11 mmHg MAP)
Brachial-to-radial gradient and capillary refill time | At baseline (after initial resuscitation). Variables will be collected only once in a cross-sectional manner.
  Correlation between brachial-to-radial gradient and capillary refill time
Brachial-to-radial gradient and lactates | At baseline (after initial resuscitation). Variables will be collected only once in a cross-sectional manner.
  Correlation between brachial-to-radial gradient and lactate concentration

CONTACTS AND LOCATIONS:
Overall Officials: Zbigniew Putowski, MD PhD, Study Chair — Center for Intensive Care and Perioperative Medicine, Jagiellonian University Medical College, Cracow, Poland
Locations (3):
- Poland (3):
  - 5 Szpital Wojskowy z Polikliniką w Krakowie, Krakow
  - Uniwersytecki Szpital w Opolu, Opole
  - Uniwersyteckie Centrum Kliniczne w Warszawie, Warsaw

IPD SHARING:
Plan to Share IPD: No